CLINICAL TRIAL: NCT02807870
Title: Early Interventions in Children With Attention Deficit/Hyperactivity Disorder: Randomized Controlled Trial Comparing Methylphenidate Parental Training in Treating Preschool Children With Attention Deficit / Hyperactivity Disorder
Brief Title: Early Interventions in Children With Attention Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Guilherme Vanoni Polanczyk, MD PhD, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 466859/2014-7
Record Dates: First submitted 2016-06-09; First posted 2016-06-21 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Preschool Child
Keywords: Parental training; Preschool age; Attention Deficit/Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Methylphenidate-psychoeducational group (Experimental): Methylphenidate treatment with a initial dosage of 0,3 mg/kg per day (weekly dosage adjustments) and weekly psychoeducational groups for parents during 8 weeks.
  Interventions: Drug: Methylphenidate; Other: Psychoeducational groups for parents
- Parental training-placebo pill (Experimental): Weekly parental training conducted by behavioral psychologists and placebo pill during 8 weeks.
  Interventions: Behavioral: Parental training; Drug: Placebo pill
- Psychoeducational group-placebo pill (Placebo Comparator): Weekly psychoeducational groups for parents and placebo pill during 8 weeks.
  Interventions: Other: Psychoeducational groups for parents; Drug: Placebo pill

INTERVENTIONS:
Drug: Methylphenidate — Methylphenidate treatment with a initial dosage of 0,3 mg/kg per day (weekly dosage adjustments).
  Arms: Methylphenidate-psychoeducational group
Behavioral: Parental training — Weekly parental training conducted by behavioral psychologists.
  Arms: Parental training-placebo pill
Other: Psychoeducational groups for parents — Weekly psychoeducational groups conducted by educators.
  Arms: Methylphenidate-psychoeducational group; Psychoeducational group-placebo pill
Drug: Placebo pill — Placebo pill during 8 weeks.
  Arms: Parental training-placebo pill; Psychoeducational group-placebo pill

SUMMARY:
Introduction: Attention deficit/hyperactivity disorder (ADHD) is one of the most prevalent mental disorders in children and is associated with important negative functional outcomes throughout development. The first signs and symptoms become apparent in preschool age. Therefore, early interventions in this population have the potential of limiting the disorder's negative impact and preventing future impairments in affected individuals. The first-choice medication for treating ADHD is methylphenidate, which has evidence of efficacy and safety in preschool children. However, non-evidence based worries and pressure from the media placed parent training as the first-line treatment for ADHD in clinical guidelines. Parent training is a behavioral intervention implemented with the parents, with weekly sessions for 8 weeks, adequate for treating ADHD dysfunctional symptoms and behaviors. However, the level of evidence for this intervention is reduced. Furthermore, the need of trained therapists in the public health system, added to the difficulties on adherence and comprehension from parents, limit its generalization and raise questions regarding its indications. Until now, no study has compared pharmacological treatment with methylphenidate to parent training in preschool children with ADHD regarding their clinical efficacy and cost-effectiveness. Moreover, no study has evaluated the impact of pharmacological intervention and psychotherapy on neurobiological mechanisms of ADHD, which is crucial for determining their impact on neurodevelopment.

Objectives: This is a double-blind randomized clinical trial that aims to evaluate the efficacy, tolerability, and acceptability of treatment with methylphenidate compared to parental training and placebo in preschool children with ADHD.

Methods: This study will be a randomized, double-blind, parallel-group, evaluating two active interventions and placebo control group. One hundred and fifty children aged 3 years and 11 months and 5 years and 11 months, diagnosed with ADHD, will be randomized to receive treatment with methylphenidate and information (50 children), parental training and treatment with placebo medication (50 children) or belong to active control group with educational information for parents and placebo treatment with no treatment (active control, 50 children). The treatment will last eight weeks, the neurobiological outcomes will be assessed before and after treatment and clinical outcomes will be assessed at weeks 0, 5 and 9. After the end of treatment, all participants will be invited to participate in a 3 years' annual follow-up. 50 children with typical development will also be evaluated in relation to neurobiological measures.

Implications: This study proposes an innovative and relevant analysis, which will enable the field to advance the knowledge of biological mechanisms related to ADHD and to treatment response. Also, the study will expand the evidence to guide early prevention strategies and early intervention.

DETAILED DESCRIPTION:
The recruitment of participants will be performed through social media divulgation, on our official website and through contact with preschools in the city of Sao Paulo. The participants that have been selected on the telephonic pre-screening are called for a diagnostic evaluation and an eligibility criteria verification performed by a child and adolescence psychiatrist and neuropsychologists. The psychiatric care and the outcomes evaluation sessions will be conducted by trained professionals, under the principal investigator's supervision.

The children will be randomized using the website randomization.com to one of the three groups: drug treatment with methylphenidate and educational information, parental training and placebo medication, or active control group with educational information and placebo medication. After the eight-week intervention, the participants can receive treatments not previously offered according to a clinical decision.

All selected participants for the clinical trial will be evaluated and accompanied by a child and adolescent psychiatrist before the study and bi-weekly until its completion. Furthermore, a blind evaluator will be responsible for the outcomes measures evaluation.

The clinical evaluator (child and adolescent psychiatrist) and the research assistant responsible for the questionnaires application will be blind towards the modality of treatment that the participant undergoes.

All of the study's evaluation protocol and monitoring is done on the platform Research Electronic Data Capture - REDCap, a software developed by Vanderbilt University - Tennessee, which is hosted in The Clinics Hospital of the University of São Paulo Medical School server. REDCap presents three main functions: a) electronic data collection; b) data management; c) study flow management. This data bank complies with the international policies of data's privacy and security on health area. In addition to the collection and storage structure, validation, auditing and data exporting tools of the system itself are also used.

The efficacy analysis will be made from treatment intention (data from all randomized patients will be included in the analysis). The outcomes (clinical measures of efficacy and tolerability) will be analyzed through mixed effects analyses, with individual models for each outcome. This model assumes that missing data occurs at random and avoids potential biases associated with the analysis only of the individuals who completed the observations or using the strategy to carry the last observation made. The model will include fixed effects for treatment (three levels), time (0, 5 and 9 weeks), time-treatment interaction and randomization effect for the participants. Effect sizes will be calculated by subtracting of the modification of each of the outcomes between the patients in the active groups versus active group control, and between both active treatments, divided by the standard deviation of the entire sample.

ELIGIBILITY:
Inclusion Criteria:

* Attention deficit hyperactivity disorder DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) diagnosis
* Score above 32 on the Swanson, Nolan, and Pelham-IV scale
* Child is registered in a school or day care center
* Children without the use of stimulants or any psychotropic in the last 30 days

Exclusion Criteria:

* Intelligence quotient <70
* The presence of clinical condition or history of neurological disorder or head trauma with conscience loss
* The presence of affective and psychotic disorders, as well as autism spectrum disorders.
* The absence of a legal representative with the capacity to understand the study objectives and the instructions related to its participation.

Ages: 47 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2016-06; Primary Completion 2019-12 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in attention deficit and hyperactivity symptoms | Baseline, after 8 weeks (post intervention) and follow-up 1, 2 and 3 years after the end of the intervention
  The child will be assessed with the Swanson, Nolan and Pelham (SNAP) scale.
Change in symptom severity | Baseline, after 8 weeks (post intervention) and follow-up 1, 2 and 3 years after the end of the intervention
  The child will be assessed by a blinded rater with the Clinical Global Impressions Scale (CGI).
Change in social and psychiatric functioning | Baseline, after 8 weeks (post intervention) and follow-up 1, 2 and 3 years after the end of the intervention
  The child will be assessed with the Children's Global Assessment Scale (CGAS).

SECONDARY OUTCOMES:
Change in executive functions | Baseline, after 8 weeks (post intervention) and follow-up 1, 2 and 3 years after the end of the intervention
  The child will be assessed with the Continuous Performance Test (CPT).
Adverse effects of the treatment | Along 8 weeks.
  The caregiver will be assessed by an adverse effects scale.
Evaluate ADHD symptoms that may influence treatment response and adherence | Baseline, after 8 weeks (post intervention) and follow-up 1, 2 and 3 years after the end of the intervention
  The caregiver will be assessed by Adult ADHD Self-Report Scale (ASRS).
Evaluate Depression symptoms that may influence treatment response and adherence | Baseline, after 8 weeks (post intervention) and follow-up 1, 2 and 3 years after the end of the intervention
  The caregiver will be assessed with Beck Depression Inventory (BDI-II)
Changes in irritability symptoms | Baseline and after 8 weeks (post intervention) and follow-up 1, 2 and 3 years after the end of the intervention
  The child will be assessed with the Affective Reactivity Index (ARI) scale.
Changes in disruptive behavior symptoms | Baseline, after 8 weeks (post intervention) and follow-up 1, 2 and 3 years after the end of the intervention
  The child will be assessed with the Multidimensional Assessment Profile of Disruptive Behavior (MAP-DB)

OTHER OUTCOMES:
Changes in Midbrain, black substance, red nucleus, median raphe, third ventricle, thalamus, anterior horn of lateral ventricles, caudate nucleus and lentiform nucleus | Baseline and after 8 weeks (post intervention).
  The child will be assessed by a transcranial ultrasound.
Changes in Expressed Emotion | Baseline and after 8 weeks (post intervention).
  The caregiver will be assessed with Five Minute Speech Sample (FMSS)
Changes in oscillatory neural connectivity | Baseline and after 8 weeks (post-intervention)
  The child will complete a battery of cognitive tasks (resting-state, Go/Nogo, emotion recognition) during electrophysiological (EEG) recording. Changes in oscillatory neural networks engaged by each task will be investigated pre- to post-intervention.
Changes in parenting behavior | Baseline and after 8 weeks (post intervention)
  Parenting behavior will be assessed by structured observation and coding performed according to the Coding System Behavior (MacMahon & Forehand, 2003).
Changes in parenting practices | Baseline and after 8 weeks (post intervention)
  Parenting practices will be assessed with the Parenting Scale (PS).
Changes in parenting practices | Baseline and after 8 weeks (post intervention)
  Parenting practices will be assessed with the Parenting Practices Scale (PPS).
Changes in parenting sense of competence | Baseline and after 8 weeks (post intervention)
  Parenting sense of competence will be assessed with the Parenting Sense of Competence Scale (PSOC).

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme V Polanczyk, Principal Investigator — University of Sao Paulo Medical School
Locations (1):
- Instituto de Psiquiatria do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sugaya LS, Salum GA, de Sousa Gurgel W, de Morais EM, Del Prette G, Pilatti CD, Dalmaso BB, Leibenluft E, Rohde LA, Polanczyk GV. Efficacy and safety of methylphenidate and behavioural parent training for children aged 3-5 years with attention-deficit hyperactivity disorder: a randomised, double-blind, placebo-controlled, and sham behavioural parent training-controlled trial. Lancet Child Adolesc Health. 2022 Dec;6(12):845-856. doi: 10.1016/S2352-4642(22)00279-6. Epub 2022 Oct 26. PMID 36306807